CLINICAL TRIAL: NCT07254247
Title: A Unique Body-Powered Terminal Device With Enhanced Grasping Capabilities for Individuals With Upper Limb Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Little Room Innovations, LLC (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R43HD115423 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (6):
- Novel Prosthetic Hook, then Control Hook (Light Spring), then Control Hook (Heavy Spring) (Experimental): In this arm, participants will first complete the tests with the Novel Prosthetic Hook and then the Control Hook with a light return spring, then the Control Hook with a heavy return spring.
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)
- Novel Prosthetic Hook, then Control Hook (Heavy Spring), then Control Hook (Light Spring) (Experimental): In this arm, participants will first complete the tests with the Novel Prosthetic Hook and then the Control Hook with a heavy return spring, then the Control Hook with a light return spring.
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)
- Control Hook (Light Spring), then Control Hook (Heavy Spring), then Novel Prosthetic Hook (Experimental): In this arm, participants will first complete the tests with the Control Hook with a light return spring, then the Control Hook with a heavy return spring, and then the Novel Prosthetic Hook.
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)
- Control Hook (Heavy Spring), then Control Hook (Light Spring), then Novel Prosthetic Hook (Experimental): In this arm, participants will first complete the tests with the Control Hook with a heavy return spring, then the Control Hook with a light return spring, and then the Novel Prosthetic Hook.
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)
- Control Hook (Light Spring), then Novel Prosthetic Hook, then Control Hook (Heavy Spring) (Experimental): In this arm, participants will first complete the tests with the Control Hook with a light return spring, then the Novel Prosthetic Hook, and then the Control Hook with a heavy return spring,
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)
- Control Hook (Heavy Spring), then Novel Prosthetic Hook, then Control Hook (Light Spring) (Experimental): In this arm, participants will first complete the tests with the the Control Hook with a heavy return spring, then Novel Prosthetic Hook, and then the Control Hook with a light return spring.
  Interventions: Device: Novel Prosthetic Hook; Device: Control Hook (Light Spring); Device: Control Hook (Heavy Spring)

INTERVENTIONS:
Device: Novel Prosthetic Hook — The Novel Prosthetic Hook is the investigational device that is being studied for its performance as an upper limb terminal device.
Device: Control Hook (Light Spring) — The Control Hook is a standard, commercially available prosthetic hook used as a comparison. In this intervention, it is configured with a light return spring.
Device: Control Hook (Heavy Spring) — The Control Hook is a standard, commercially available prosthetic hook used as a comparison. In this intervention, it is configured with a heavy return spring.

SUMMARY:
We have developed a novel terminal device for a prosthetic arm that eliminates the functional tradeoffs seen in body-powered voluntary open devices. The primary goal of this study is to validate the performance of the device against the commercial state-of-the-art in upper limb terminal devices.

ELIGIBILITY:
Inclusion Criteria:

Are between the ages of 18-80 Are proficient in English Able to demonstrate proper functioning and safety of the terminal device

Exclusion Criteria:

Have visual or mental impairments Have history of neurological or musculoskeletal disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Modified SHAP Average Completion Time | through study completion, an average of 1 day
  This is the average task completion time across all tasks performed in a modified version of the Southampton Hand Assessment Protocol (SHAP). The SHAP has been modified in this study to include only the relevant assessments to the prosthetic hooks being tested. A lower average score indicates better performance.

SECONDARY OUTCOMES:
Clothespin Relocation Task Average Time | through study completion, an average of 1 day
  This is a functional hand assessment that measures the time it takes to reposition clothespins of differing stiffnesses. Lower completion times indicate better performance.
Borg Rating of Perceived Exertion (RPE) | through study completion, an average of 1 day
  This is a scale of 0 to 10 with 0 indicated by the participate as a measure of how difficult a task is.
NASA Task Load Index | through study completion, an average of 1 day
  The NASA Task Load Index method assesses work load. The aggregate score reported scales from 0 to 100, where 100 indicates the maximum (hardest) workload.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided